CLINICAL TRIAL: NCT06136663
Title: A Prospective Cohort Survey on Prevalence and Risk Factors for Persistent Postsurgical Pain After the Open Reduction and Internal Fixation of the Lower Limbs
Brief Title: Prevalence and Risk Factors for Postsurgical Pain After the Open Reduction and Internal Fixation of Lower Limbs.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XZXY-LK-20230530-085
Record Dates: First submitted 2023-10-31; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Chronic Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pain-free control subjects: Patients with no postoperative chronic pain after open reduction and internal fixation of lower limb fractures.
- Patients with chronic postsurgical pain: Patients with postsurgical chronic pain after open reduction and internal fixation of lower limb fractures.

SUMMARY:
The objective of this study is to specify the demographic and medical factors that most likely constitute a risk of developing CPSP in the patients with lower limb.

DETAILED DESCRIPTION:
Chronic pain,one of the most frequent causes for patients to seek medical care,is a recognized health problem.Chronic postsurgical pain (CPSP), commonly defined as pain that develops after a surgical procedure and persists at least 3 months, constitutes a widely underdiagnosed and often poorly treated medical problem affecting 10-50% of all postsurgical patients. According to the reports,in the United States alone,1.9 million persons abused or were dependent on prescription opioid analgesics for chronic pain in 2013,contributing to one of the worst public health crises the developed world has recently faced.Here,open reduction and internal fixation（ORIF） of lower limb fractures ,what the investigators focus, is a common surgical procedure in orthopedics and microscopic hand and foot surgery.The removal of the intramedullary nail can relieve anterior knee pain, but in a substantial number of patients, pain persists after nail removal.The most painful daily activities are kneeling and squatting.Therefore, it is increasingly important and urgent to solve the postoperative chronic pain of patients with lower extremity fractures surgery.

The underlying biology of chronic postoperative pain and genetic heritability is complex and not yet fully understood . A common feature of CPSP is that the painful sensations change from the familiar acute postoperative pain to a complex pain syndrome with nonaplastic characteristics，neuropathic characteristics, or both. Preclinical studies have revealed that neuroinflammation is one of pathological hallmarks of CPSP. The transition from acute to chronic pain starts early within the first 2 weeks after nonaplastic by peripheral and central inflammatory processes and activation of spinal glial cells.Repetitive nociception resulting from prolonged inflammatory and neuropathic responses to noxious stimuli causes a cascade of biochemical and structural changes to various pain pathways resulting in sensitization of the peripheral and central nervous system（CNS）. Cytokines and neurotrophic factors have been identified as pivotal mediators involved in neuroimmune activation pathways and cascades in various preclinical chronic pain models.

Although lower limb fracture is one of the most frequently reported triggering CPSP events, few large-scale studies have shown the occurrence of and factors associated with it.The objectives of investigators are to specify the demographic and medical factors that most likely constitute a risk of developing CPSP and to search for potential interventions to reduce the occurrence of CPSP in these limb fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Underwent surgical repair including fracture of the lower leg, fracture of the foot and fractures involving multiple regions of the lower limbs.

Exclusion Criteria:

* Refusing to participate in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to trauma center for lower fracture (femur, tibia, patella, or foot/ankle) requiring open-reduction internal fixation were screened for inclusion between January 2020 and March 2023. Demographic questions are completed at the time of consent, and the mechanism of injury, primary injury location, body mass index, blood and urine assessments are extracted from each individual's medical record. Additionally, at 3 months each participant was asked whether they had developed chronic pain and completed a validated measure of self-reported pain intensity.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative chronic pain：pain score | Through study completion, an average of 1 year
  1. Postoperative chronic pain assessed by the Numerical Rating Scale (NRS). Pain score >=3 at operational areas (minimum 0, maximum 10, higher score indicates greater pain).
  2. Pain developed after a surgical procedure or increased in intensity after the surgical procedure.
  3. Pain should be of at least 3 months duration with a significant negative effect on the quality of life.
  4. Pain is a continuation of acute postoperative pain or may develop after an asymptomatic period and pain is localized to the surgical field or to a referred area (eg, innervation territory, referred dermatome for visceral surgery).
  5. Other possible causes for the pain have been excluded (eg, infection, cancer recurrence)
Perioperative inflammatory state | Up to 10 days
  The inflammatory factors，C-reactive protein（CRP）, white blood cell count, and lymphocyte ratio of the subjects were counted.
Lifestyle and behaviour of the subjects | Baseline
  Through the electronic medical record system and telephone follow-up, to understand whether there is a history of smoking, drinking, physical activity.
Preoperative complications of the participants | Baseline
  Including cardiovascular and cerebrovascular diseases (such as hypertension, coronary heart disease), respiratory diseases (such as chronic obstructive pulmonary disease), endocrine system diseases (such as diabetes, hyperthyroidism) and so on.
Medical interventions history | Up to 10 days
  The use of the analgesic drugs， including the past and this perioperative period
Surgery details | Baseline
  Including specific surgical site (femur, tibia or fibula or multiple injuries) ，the time of operation, the amount of bleeding during operation，etc.
Anesthesia during surgery | Baseline
  The types of anesthesia (general anesthesia, spinal anesthesia and whether to use nerve block, etc. )
Age | Baseline
  The age of each subject in the operating room was counted.
Body mass index (BMI) | Baseline
  The BMI of each subject in the operating room was counted and compared.
Gender | Baseline
  The gender ratio of the CPSP group and pain-free group was recorded and compared.
Cultural background | Baseline
  Record the highest academic qualifications of the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

REFERENCES:
- [Background] Scholz J, Finnerup NB, Attal N, Aziz Q, Baron R, Bennett MI, Benoliel R, Cohen M, Cruccu G, Davis KD, Evers S, First M, Giamberardino MA, Hansson P, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Nurmikko T, Perrot S, Raja SN, Rice ASC, Rowbotham MC, Schug S, Simpson DM, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ, Barke A, Rief W, Treede RD; Classification Committee of the Neuropathic Pain Special Interest Group (NeuPSIG). The IASP classification of chronic pain for ICD-11: chronic neuropathic pain. Pain. 2019 Jan;160(1):53-59. doi: 10.1097/j.pain.0000000000001365. PMID 30586071
- [Background] van Ransbeeck A, Budilivski A, Spahn DR, Macrea L, Giuliani F, Maurer K. Pain Assessment Discrepancies: A Cross-Sectional Study Highlights the Amount of Underrated Pain. Pain Pract. 2018 Mar;18(3):360-367. doi: 10.1111/papr.12612. Epub 2017 Sep 20. PMID 28707777
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Clay FJ, Watson WL, Newstead SV, McClure RJ. A systematic review of early prognostic factors for persisting pain following acute orthopedic trauma. Pain Res Manag. 2012 Jan-Feb;17(1):35-44. doi: 10.1155/2012/935194. PMID 22518366
- [Background] Friesgaard KD, Gromov K, Knudsen LF, Brix M, Troelsen A, Nikolajsen L. Persistent pain is common 1 year after ankle and wrist fracture surgery: a register-based questionnaire study. Br J Anaesth. 2016 May;116(5):655-61. doi: 10.1093/bja/aew069. PMID 27106969
- [Background] Leliveld MS, Van Lieshout EMM, Polinder S, Verhofstad MHJ; TRAVEL Study Investigators. Effect of Transverse Versus Longitudinal Incisions on Anterior Knee Pain After Tibial Nailing (TRAVEL): A Multicenter Randomized Trial with 1-Year Follow-up. J Bone Joint Surg Am. 2022 Dec 21;104(24):2160-2169. doi: 10.2106/JBJS.22.00389. Epub 2022 Oct 25. PMID 36367768
- [Background] Wyss-Coray T, Mucke L. Inflammation in neurodegenerative disease--a double-edged sword. Neuron. 2002 Aug 1;35(3):419-32. doi: 10.1016/s0896-6273(02)00794-8. PMID 12165466
- [Background] Fitzcharles MA, Cohen SP, Clauw DJ, Littlejohn G, Usui C, Hauser W. Nociplastic pain: towards an understanding of prevalent pain conditions. Lancet. 2021 May 29;397(10289):2098-2110. doi: 10.1016/S0140-6736(21)00392-5. PMID 34062144
- [Background] Hankerd K, McDonough KE, Wang J, Tang SJ, Chung JM, La JH. Postinjury stimulation triggers a transition to nociplastic pain in mice. Pain. 2022 Mar 1;163(3):461-473. doi: 10.1097/j.pain.0000000000002366. PMID 34285154
- [Background] Lavand'homme P. Transition from acute to chronic pain after surgery. Pain. 2017 Apr;158 Suppl 1:S50-S54. doi: 10.1097/j.pain.0000000000000809. No abstract available. PMID 28134653
- [Result] Rees S, Tutton E, Achten J, Bruce J, Costa ML. Patient experience of long-term recovery after open fracture of the lower limb: a qualitative study using interviews in a community setting. BMJ Open. 2019 Oct 9;9(10):e031261. doi: 10.1136/bmjopen-2019-031261. PMID 31601595
- [Result] Van Wyngaarden JJ, Archer KR, Pennings JS, Matuszewski PE, Noehren B. Psychosocial Predictors of Chronic Pain 12 Months After Surgical Fixation for Lower Extremity Fracture: A Prospective Study. Phys Ther. 2022 Oct 6;102(10):pzac101. doi: 10.1093/ptj/pzac101. PMID 35926071